CLINICAL TRIAL: NCT00022308
Title: Phase I Trial of Radical Thoracic Radiation, Weekly CPT-11 (Irinotecan) and Cisplatin in Locally Advanced Non-Small Cell Lung Carcinoma
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068803; P30CA006927 (NIH); FCCC-98020; NCI-G01-1995
Record Dates: First submitted 2001-08-10; First posted 2004-02-27 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Irinotecan; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients who have locally advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of irinotecan when administered with cisplatin and radiotherapy in patients with locally advanced non-small cell lung carcinoma. II. Determine the toxic effects, especially acute and long-term esophagitis and pneumonitis, of this regimen in these patients. III. Determine the response rate, duration to progression, and sites of relapse in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of irinotecan. Patients receive irinotecan IV over 90 minutes and cisplatin over 1 hour on day 1. Patients also undergo radiotherapy once daily on days 1-5. Treatment repeats every 7 days for 7 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients are followed every 2 months for 1 year, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 3-27 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) Stage IIIB or bulky stage IIIA not amenable to surgical resection Medically inoperable stage II or non-bulky stage IIIA Locally recurrent disease following surgery that is not amenable to further surgical resection No small cell carcinoma or mixed cytology No disease beyond radiation portal (T4 tumors with documented multifocal malignant pleural involvement or extension of supraclavicular nodal disease to cervical chain) No pleural effusion Pleural effusions visible on CT scan but not on chest x-ray that are inaccessible to thoracentesis or are cytologically negative are allowed Ineligible for enrollment on protocol RTOG 93-09

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL No known Gilbert's disease Renal: Creatinine no greater than 1.5 mg/dL Calcium less than 12.0 mg/dL Cardiovascular: No symptomatic cardiovascular disease No active angina No congestive heart failure requiring active therapy No uncontrolled arrhythmias No myocardial infarction within the past 6 months Pulmonary: FEV1 at least 1.0 L unless cleared by radiation oncologist Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception for 3 months before study, during study, and for 3 months after study HIV negative No other concurrent active or invasive malignancy except nonmelanoma skin cancer Less than 10% unintended weight loss within 3 months of diagnosis No other concurrent medical condition that would preclude study No social situation or psychiatric disorder that would preclude study No active or uncontrolled infection No history of seizures No uncontrolled diabetes mellitus (random blood sugar at least 250 mg/dL)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for NSCLC No prior irinotecan or topotecan Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for NSCLC No prior radiotherapy to the chest Surgery: See Disease Characteristics Other: No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (8):
- United States (8):
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania

REFERENCES:
- [Result] Langer CJ, Somer R, Litwin S, Feigenberg S, Movsas B, Maiale C, Sherman E, Millenson M, Nicoloau N, Huang C, Treat J. Phase I study of radical thoracic radiation, weekly irinotecan, and cisplatin in locally advanced non-small cell lung carcinoma. J Thorac Oncol. 2007 Mar;2(3):203-9. doi: 10.1097/JTO.0b013e318031cd3c. PMID 17410043